CLINICAL TRIAL: NCT00630396
Title: Minocycline to Improve Neurologic Outcome in Stroke (MINOS)
Brief Title: Study of a Neuroprotective Drug to Limit the Extent of Damage From an Ischemic Stroke
Acronym: MINOS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: David Hess, MD (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); University of Kentucky (Other); Oregon Health and Science University (Other)
Responsible Party: Sponsor-Investigator, David Hess, MD, Professor and Chairman, Augusta University
Organization: Augusta University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R01NS055728-01A1 (NIH); 07-02-202 (Other: GHSU Human Assurance Committee number)
Record Dates: First submitted 2008-02-28; First posted 2008-03-07 (Estimated); Results first posted 2012-01-13 (Estimated); Last update posted 2012-01-13 (Estimated); Status verified 2011-12

CONDITIONS: Stroke, Acute
Keywords: stroke; ischemic; neuroprotection; minocycline; tissue plasminogen activator (tPA); biomarkers; pharmacokinetics; antiapoptotic; anti-inflammatory; treatment; matrix metalloproteinase-9 (MMP-9); thrombolysis; Minocycline to Improve Neurologic Outcome in Stroke (MINOS); cerebrovascular stroke; cerebrovascular accident; cerebral stroke; cerebrovascular accident (CVA)
MeSH Terms: conditions — Stroke; Ischemia; cyclopia sequence | interventions — Minocycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Minocycline — Dose level 1 = 3mg/kg intravenous (IV) initial dose, followed by 1.5mg/kg every 12 hours times 5 more doses.
  Dose level 2 = 4.5mg/kg intravenous (IV) initial dose, followed by 2.25mg/kg every 12 hours times 5 more doses.
  Dose level 3 = 6 mg/kg intravenous (IV) initial dose, followed by 3 mg/kg every 12 hours times 5 more doses.
  Dose level 4 = 10 mg/kg intravenous (IV) initial dose, followed by 5 mg/kg every 12 hours times 5 more doses
  Other Names: Minomycin; Minocycline hydrochloride; Minocycline hydrochloride injection; Minomycin Intravenous (for drip use); Minomycin Intravenous; MINO

SUMMARY:
The primary aim of this study is to find out which of 4 different doses of minocycline are safe and well tolerated so that we will know the optimal dose to test in future patients.

DETAILED DESCRIPTION:
Minocycline is a widely used antibiotic and is approved by the Food and Drug Administration (FDA) for treatment of infections and acne. However, doctors do not know whether minocycline will work in stroke patients. Its use in stroke patients is experimental. There is a lot of information from experimental stroke studies in animals that minocycline lessens the damage from a stroke and the animals recover better. Since minocycline is generally a very safe drug in humans and does not have a lot of side effects, investigators at Georgia Health Sciences University (formerly the Medical College of Georgia) believe that it might be a safe and effective drug to improve the outcome in patients with stroke.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years of age
* acute onset focal neurologic deficit consistent with acute ischemic stroke, or computed tomographic scan consistent with acute cerebral ischemia
* onset of symptoms less than 6 hours
* measurable neurologic deficit (National Institutes of Health [NIH] Stroke Scale >/= 1)

Exclusion Criteria:

* allergy to tetracycline antibiotics
* women of child-bearing potential
* known hepatic and/or renal insufficiency
* Thrombocytopenia
* history of intolerance to minocycline
* dizziness at the time of stroke or in the past month (by self-report)
* aphasia likely to interfere with patients ability to report adverse effects
* previous functional disability
* stuporous or comatose
* presence of another serious illness likely to confound the study
* unlikely to be available for 90 day follow-up
* severe stroke (National Institutes of Health [NIH] Stroke Scale >22)
* undergoing an interventional neuro-radiological intervention in first 12 hour

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-05; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David C Hess, MD, Principal Investigator — Augusta University
Locations (2):
- United States (2):
  - University of Kentucky, Lexington, Kentucky
  - Oregon Health & Science University, Portland, Oregon

REFERENCES:
- [Result] Fagan SC, Waller JL, Nichols FT, Edwards DJ, Pettigrew LC, Clark WM, Hall CE, Switzer JA, Ergul A, Hess DC. Minocycline to improve neurologic outcome in stroke (MINOS): a dose-finding study. Stroke. 2010 Oct;41(10):2283-7. doi: 10.1161/STROKEAHA.110.582601. Epub 2010 Aug 12. PMID 20705929

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred from June 3, 2008 to October 10, 2009. The study was completed ahead of schedule. Study subjects were enrolled in each recruiting centers' Emergency Department or stroke intensive care unit. Many subjects came as transfers from rural or outside hospitals to one of the enrolling centers for further care and study participation.
Pre-assignment Details: Potential patients that met all of the inclusion criteria, did not meet any of the exclusion criteria, and were willing to participate were enrolled in the study. All study subjects were given one of the four doses of minocycline. The dose of minocycline given was assigned by a computer program.
Groups:
- Minocycline: All 60 participants were treated with minocycline. 11 participants were treated at 3mg/kg, 4 were treated at 4.5mg/kg, 4 were treated at 6mg/kg, and 41 were treated at 10mg/kg.
Period: Overall Study
Arm/Group | Minocycline
Started | 60
Completed | 53
Not Completed | 7
Not completed — Death | 4
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Arm/Group | Minocycline
Number analyzed (Participants) | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 30
Age Continuous [Mean (Standard Deviation); unit: years]
  Overall age | 65 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 32
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 50
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 60
Weight [Mean (Standard Deviation); unit: Kg] | 81.6 (21.6)
Subjects receiving t-PA then minocycline [Number; unit: Participants] — Patients that received tissue plasminogen activator (tPA) were also eligible for the MINOS trial. Once tPA had finished infusing, the research team would commence with the study drug infusion.
  Participants
    Total amount of subjects that received t-PA | 36
    Total amount of subjects that did not receive t-PA | 24
NIH Stroke Scale at baseline [Mean (Standard Deviation); unit: Units on a scale] — The National Institutes of Health (NIH) Stroke Scale was designed to assess, score, and reliably communicate the level of impairment in a stroke patient. The maximum score is a 42, and the minimum score is a 0. A 42 represents the most severe stroke as scored by the NIH Stroke Scale.
  Units on a scale | 8.7 (5.8)
Symptom onset to study drug infusion time [Mean (Standard Deviation); unit: minutes] — This is the average time from when the patient was "last known to be normal" to the moment the study drug began infusing intravenously.
  minutes | 307.4 (50.0)

OUTCOME MEASURES:

1. Primary Outcome: Maximally Tolerated Dose of IV Minocycline
Description: Investigators closely monitored each subject for evidence of minocycline intolerance. All adverse events were immediately reported for a decision whether to discontinue the study medication and/or reduce the dose. A computer program was used to determine the maximum tolerated dose. After entering information regarding doses and expected toxicities, results for each subject as they were collected were entered. The computer program informed as to (de)escalation, or maintenance of the same dose in the subsequent cohort of enrolled patients.
Time Frame: 3 days
Measure: Number; unit: mg/kg
Arm/Group | Minocycline
Number analyzed (Participants) | 60
mg/kg | 10

2. Secondary Outcome: Half-life of IV Minocycline
Description: In eligible patients enrolled at Georgia Health Sciences University, blood samples were drawn for quantification of minocycline serum concentrations. This enabled the study team to determine the half life of the study drug.
Time Frame: For each subject blood samples were drawn before dose #1 and one hour after starting dose #1. Additional blood was drawn 1, 6, 12, 24, 48, and 72 hours after starting dose #6, which lasted approximately 6 days.
Measure: Mean (Standard Error); unit: hours
Units Other Than Participants: blood samples
Arm/Group | Minocycline
Number analyzed (Participants) | 22
Number analyzed (blood samples) | 176
hours | 23.8 (1.9)

3. Secondary Outcome: 90 Day Modified Rankin Scale Score
Description: The modified Rankin Scale (mRS) was performed in person at the 90 day clinic follow-up appointment. The modified Rankin Scale is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke. The scale runs from 0-6. 0 represents no symptoms. 1 represents no significant disability. 2 represents slight disability. 3 represents moderate disability. 4 represents moderately severe disability. 5 represents severe disability. 6 represents death.
Time Frame: 3 months
Measure: Number; unit: Participants
Arm/Group | Minocycline
Number analyzed (Participants) | 60
Participants
  90 day mRS score of 0 overall | 15
  90 day mRS score of 1 overall | 15
  90 day mRS score of 2 overall | 9
  90 day mRS score of 3 overall | 11
  90 day mRS score of 4 overall | 2
  90 day mRS score of 5 overall | 3
  90 day mRS score of 6 overall | 5

ADVERSE EVENTS:
Time Frame: Adverse Events were collected for one year and seven months. This time period started when the first subject was enrolled and lasted until the 90 day follow-up was completed for the last subject enrolled.
Description: Investigators closely monitored each patient for evidence of study drug intolerance, particularly focusing on dizziness, gastrointestinal complaints, and infusion reactions.
Arm/Group | Minocycline
Serious Adverse Events (participants affected / at risk) | 29/60
Other Adverse Events (participants affected / at risk) | 50/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Minocycline (N=60)
Death (Nervous system disorders) | 5 (5) — Five individuals died during the study. Three occurred during hospitalization(all three were attributed to the patient's underlying illness). The other two deaths after discharge were from gastric cancer and worsening congestive heart failure.
Transient Ischemic Attack (Nervous system disorders) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 3 (3)
Acute Ischemic Stroke (Nervous system disorders) | 3 (3)
Worsening hallucinations and agitation (Nervous system disorders) | 1 (1)
Congestive Heart Failure exacerbation (Cardiac disorders) | 1 (1)
Rule out myocardial infarction (chest pain, nausea, shortness of breath) (Cardiac disorders) | 1 (1) — Subject complained of chest pain at home. Subject was hospitalized. Cardiac enzymes and chest x-ray were negative. Chest pain resolved, and myocardial infarction was ruled out.
Congestive Heart Failure (Cardiac disorders) | 1 (1)
Neuroworsening (Nervous system disorders) | 3 (3) — Neuroworsening is an increase in the severity of a subject's stroke (defined as an increase in a subjects National Institutes of Health Stroke Scale by 4 or more points).
Left hip fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Pulmonary emboli secondary to left lower extremity deep vein thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Carotid endarterectomy (Surgical and medical procedures) | 1 (1)
Rule out pneumonia (Infections and infestations) | 1 (1) — Subject hospitalized and thought to have left lower lobe pneumonia based on chest x-ray. He received 1 dose of 2 different antibiotics. Subject improved; however, subject not thought to have pneumonia. Subject was discharged home without antibiotics.
Scrotal edema (Reproductive system and breast disorders) | 1 (1)
Stomach cancer (Gastrointestinal disorders) | 1 (1)
Paroxysmal atrial fibrillation (Cardiac disorders) | 1 (1)
Depression/suicide attempt (Psychiatric disorders) | 1 (1)
Hypotension (Renal and urinary disorders) | 1 (1)
Intracerebral Hemorrhage (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Minocycline (N=60)
Hemorrhagic transformation (Nervous system disorders) | 3 (3)
Neurological worsening (Nervous system disorders) | 3 (3)
GI Symptoms (Gastrointestinal disorders) | 12 (22) — Nausea, vomiting, diarrhea, stomach pain, epigastric pain, abdominal pain, excessive belching, worsening dyspepsia
Skin reactions (Skin and subcutaneous tissue disorders) | 13 (17) — Phlebitis (0), Burning at the IV site during infusion, Stage I & II skin breakdown, rash and bruising.
Urinary Tract Infection (Infections and infestations) | 3 (3)
Atrial Fibrillation (Cardiac disorders) | 3 (3)
Elevated liver enzymes (Renal and urinary disorders) | 4 (4) — Elevated liver enzymes (2), elevated LFTs (1), and hepatic toxicity (1).
Reduced platelet count (Blood and lymphatic system disorders) | 4 (4)
Headache (Nervous system disorders) | 15 (15) — There were 13 complaints of headache and 2 complaints of worsening of headache.
Vertigo (Nervous system disorders) | 3 (4) — Disequilibrium (1) and dizziness (3)
Hypotension (Renal and urinary disorders) | 4 (4)
Pain (General disorders) | 10 (13) — Complaints of pain occurred in the: shoulder, neck, foot, knee, back, hand, leg, left lower extremity and penis (1).
Chest pain (Cardiac disorders) | 4 (4)
Tachycardia (Cardiac disorders) | 3 (3)
Aspiration pneumonia (Infections and infestations) | 3 (3)
Edema (General disorders) | 3 (4) — Peripheral edema (1 case); mild pulmonary edema (1 case); bilateral upper extremity edema (1 case); lower extremity edema (1 case)

LIMITATIONS AND CAVEATS:
Some statistical tests could not be performed due to small sample size in the 4.5 and 6mg/kg dose tiers.

The modified continual reassessment method (CRM) failed to identify the maximum tolerated dose of intravenous minocycline.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No